CLINICAL TRIAL: NCT06888570
Title: Childhood Obesity is a Global Health Issue, Especially in Children With Trisomy 21 (T21), Who Face Higher Risks of Non-alcoholic Fatty Liver Disease (NAFLD). Early Detection Using Non-invasive Tools Like Liver Elastography is Key. Evaluating Dietary Patterns With the 24-hour Food Recall and KIDMED Helps Guide Personalized Interventions
Brief Title: Relationship Between Eating Patterns, Body Composition and the Detection of Fatty Liver in Children and Adolescents With Trisomy 21: LiverTy Project
Acronym: LiverTy
Status: Enrolling by invitation | Type: Observational
Sponsor: IMDEA Food (Other)
Responsible Party: Principal Investigator, Lorena Lopez Lora, Nurse and Nutricionist, IMDEA Food
Other Study IDs: IMD: PI-070
Record Dates: First submitted 2025-02-28; First posted 2025-03-21 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Obesity Prevention; Pediatric Obesity; Trisomy 21; Down Syndrome (Trisomy 21); Elastography; Nutrition Assessment; Liver Diseases; Non Alcoholic Fatty Liver Disease; Body Composition
Keywords: Fibroscan; Fatty liver disease; Body composition; Trisomy 21; Down Syndrome; KIDMED questionnaire; 24-hour dietary recall; Non-invasive liver assessment; Non Alcoholic Fatty Liver Diseases; Obesity prevention; Children; Adolescents
MeSH Terms: conditions — Pediatric Obesity; Down Syndrome; Liver Diseases; Non-alcoholic Fatty Liver Disease | interventions — Population Control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group.: Children and adolescents (ages 5-22) with Down syndrome (T21) who may have or not have NAFLD.
  Interventions: Other: To evaluate fat liver content in the cases/controls population.
- Control group.: Children and adolescents (ages 5-22) without Down syndrome (T21) who may have or not have NAFLD.
  Interventions: Other: To evaluate fat liver content in the cases/controls population.

INTERVENTIONS:
Other: To evaluate fat liver content in the cases/controls population. — The studied population includes participants aged 5-22 years old with/without T21 Down Syndrome.

SUMMARY:
Childhood obesity is a growing public health issue affecting millions of children worldwide, increasing the risk of metabolic and cardiovascular diseases in adulthood. This problem is particularly concerning in children and adolescents with Down syndrome (trisomy 21, T21), who have a higher predisposition to fat accumulation due to genetic, metabolic, and behavioral factors. However, assessing their nutritional status and body composition is challenging, as conventional tools such as body mass index (BMI) may not accurately reflect adiposity in this population.

One of the most severe risks associated with obesity in children with T21 is non-alcoholic fatty liver disease (NAFLD). This condition is characterized by fat accumulation in the liver without significant alcohol consumption and is closely linked to insulin resistance, dyslipidemia, and pro-inflammatory states. If not detected early, NAFLD can progress to more severe liver diseases such as fibrosis or cirrhosis. In individuals with T21, the prevalence of NAFLD may be underestimated due to the difficulty in properly assessing body composition and metabolism.

Since NAFLD diagnosis traditionally requires invasive procedures such as liver biopsy, this study proposes using non-invasive techniques, such as liver elastography, to assess liver health in children and adolescents with T21. Additionally, dietary habits will be analyzed using standardized tools to establish the relationship between nutrition, body composition, and NAFLD risk in this population.

Study Hypothesis:

The main hypothesis is that obesity and inadequate dietary patterns increase the risk of NAFLD in our participants with T21. The investigators also believe that liver elastography will enable the early detection of fat accumulation in the liver and other signs of liver disease, facilitating timely intervention.

Study Objectives:

The primary objective of this study is to evaluate the presence and severity of NAFLD in children and adolescents with T21 using non-invasive diagnostic techniques and nutritional assessment methods.

Specifically, the study will analyze:

* Liver health: Measurement of liver fat and stiffness using elastography. Body composition: Anthropometric evaluation and adiposity analysis. Dietary habits: 24-hour food recall and KIDMED questionnaire to assess adherence to the Mediterranean diet.
* Relationship between obesity and NAFLD: Identification of metabolic and behavioral risk factors.

DETAILED DESCRIPTION:
1. Study Design

   This is an observational cross-sectional study in which participants with T21, with and without obesity, will be evaluated without direct therapeutic intervention.
2. Registration and Evaluation Procedures

   2.1 Clinical Assessments
   * Liver Elastography: Assessment of liver stiffness using FibroScan. Hepatic elastography is a non-invasive imaging technique used to assess liver stiffness and fat content, which correlates with liver fibrosis. It is particularly useful in pediatric populations for evaluating liver diseases such as non-alcoholic fatty liver disease (NAFLD), viral hepatitis, and other chronic liver conditions. FibroScan measures ultrasound signal attenuation due to liver fat content. Higher values (db/m) indicate more fat deposition.
   * Anthropometric Measurements: Weight, height, body mass index (BMI), abdominal circumference.
   * Body composition parameters measured by bioimpedance:

   Adipose tissue %, muscle mass (kg) and visceral fat index.

   2.2. Nutritional Evaluation:
   * 24-hour dietary recall. To estimate nutrient consumption, dietary intake from the 24-hour dietary recall will be converted given the use of nutritional composition tables and validated food composition software (DIAL).
   * KIDMED questionnaire for adherence to the Mediterranean diet.

   The KIDMED (Mediterranean Diet Quality Index) questionnaire is a widely used tool to assess adherence to the Mediterranean diet among children and adolescents. It consists of 16 items that evaluate various dietary habits. Each item is scored as follows:

   Positive connotation items (reflecting healthy Mediterranean dietary habits): Each receives a score of +1.

   Negative connotation items (indicating departure from Mediterranean dietary principles): Each receives a score of -1.

   The total KIDMED score ranges from -4 to 12. Based on the total score, adherence to the Mediterranean diet is categorized into three levels:

   High adherence: Scores of ≥8. Medium adherence: Scores between 4 and 7. Low adherence: Scores of ≤3.
3. Quality Assurance Plan

   Electronic data management system with automatic validations to prevent data entry errors.
4. Sample Size Evaluation

   It is estimated that a sample of 17 participants with T21 and 17 participants in the control group reaches 80% statistical power in detecting significant differences in the detection of fatty liver.
5. Statistical Analysis Plan

   * Descriptive statistics will be used to characterize the sample.
   * Correlation tests and logistic regression will be performed to assess the relationship between NAFLD and metabolic factors.
   * Analysis of variance (ANOVA) will be used to compare parameters among subgroups.
6. Ethical and Safety Considerations

   * Approval from the Research Ethics Committee.
   * Data management in compliance with the General Data Protection Regulation (GDPR).

This protocol will allow us to evaluate the relationship between obesity, dietary patterns, and NAFLD in children with T21, providing key information for future preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Children (5-10 years), and adolescents (11-19) andyoung adults (20-22 years) of bothSexes
* 5 to 22 years old
* Diagnosis of trisomy 21 or other intellectual disability of genetic origin for the group of the cases.
* BMI: 17-40 Kg/m2
* Signing of the informed consent by the parents or guardians.

Exclusion Criteria:

* Not meeting the inclusion criteria
* Have previous liver pathology.
* Be under any medical treatment that
* Modify composition parameters Body: GLP-1 analogues and derivatives.

Ages: 5 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be selected who are patients at the Jerome Lejeune Foundation center or students in special education centers who wish to participate. For the control group, dissemination will be carried out among workers with children of the required age range.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Liver fat content. | 3 months.
  To estimate liver fat content with hepatic elastography (FibroScan), CAP measurement will be used. Control population CAP value would range between 160-184 db/m and cases ≥ 184 db/m.

SECONDARY OUTCOMES:
Body weight. | 3 months.
  Body weight (kg) will be assessed with a calibrated scale with the purpose of obtaining descriptive data of both populations, cases and controls.
Height. | 3 months.
  Height (cm) will be assessed with a calibrated stadiometer with the purpose of obtaining descriptive data of both populations, cases and controls.
Body Mass Index. | 3 months.
  Body Mass Index (kg/m*2) will be calculated with the body weight and height.
Waist circumference. | 3 months.
  Waist circumference (cm) will be assessed with a measuring tape with the purpose of obtaining descriptive data of both populations, cases and controls.
Adipose tissue (%). | 3 months.
  Adipose tissue (%) will be estimated with bioimpedance with a calibrated TANITA with the purpose of obtaining descriptive data of both populations, cases and controls.
Visceral fat index. | 3 months.
  Visceral fat index will be estimated with bioimpedance with a calibrated TANITA with the purpose of obtaining descriptive data of both populations, cases and controls.
Muscle mass. | 3 months.
  Muscle mass (kg) will be estimated with bioimpedance with a calibrated TANITA with the purpose of obtaining descriptive data of both populations, cases and controls.
24-hour dietary quality evaluation. | 3 months.
  24-hour dietary quality will be assessed with a validated 24-h recall food questionnaire in both populations, cases and controls.
Mediterranean diet adherence. | 3 months.
  Mediterranean diet adherence will be assessed with a validated mediterranean food questionnaire for pediatric population (KIDMED) in both, cases and controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Jerome Lejeune, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Relevant data obtained on the relationship of fatty liver in the studied population

REFERENCES:
- [Background] Altavilla C, Caballero-Perez P. An update of the KIDMED questionnaire, a Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2019 Oct;22(14):2543-2547. doi: 10.1017/S1368980019001058. Epub 2019 May 31. PMID 31146796
- [Background] Hewawitharana SC, Thompson FE, Loria CM, Strauss W, Nagaraja J, Ritchie L, Webb KL. Comparison of the NHANES dietary screener questionnaire to the Automated Self-Administered 24-Hour Recall for Children in the Healthy Communities Study. Nutr J. 2018 Nov 27;17(1):111. doi: 10.1186/s12937-018-0415-1. PMID 30482218
- [Background] Arsoy HA, Kara O, Keskin M. The evaluation of non-alcoholic fatty liver disease in children with obesity with vibration-controlled transient elastography. J Clin Ultrasound. 2024 Jul-Aug;52(6):723-730. doi: 10.1002/jcu.23698. Epub 2024 Apr 18. PMID 38635340
- [Background] Castera L, Friedrich-Rust M, Loomba R. Noninvasive Assessment of Liver Disease in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2019 Apr;156(5):1264-1281.e4. doi: 10.1053/j.gastro.2018.12.036. Epub 2019 Jan 18. PMID 30660725
- [Background] Hielscher L, Irvine K, Ludlow AK, Rogers S, Mengoni SE. A Scoping Review of the Complementary Feeding Practices and Early Eating Experiences of Children With Down Syndrome. J Pediatr Psychol. 2023 Nov 16;48(11):914-930. doi: 10.1093/jpepsy/jsad060. PMID 37738668
- [Background] Vos MB, Abrams SH, Barlow SE, Caprio S, Daniels SR, Kohli R, Mouzaki M, Sathya P, Schwimmer JB, Sundaram SS, Xanthakos SA. NASPGHAN Clinical Practice Guideline for the Diagnosis and Treatment of Nonalcoholic Fatty Liver Disease in Children: Recommendations from the Expert Committee on NAFLD (ECON) and the North American Society of Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN). J Pediatr Gastroenterol Nutr. 2017 Feb;64(2):319-334. doi: 10.1097/MPG.0000000000001482. PMID 28107283
- [Background] Goldner D, Lavine JE. Nonalcoholic Fatty Liver Disease in Children: Unique Considerations and Challenges. Gastroenterology. 2020 May;158(7):1967-1983.e1. doi: 10.1053/j.gastro.2020.01.048. Epub 2020 Mar 20. PMID 32201176
- [Background] Bertapelli F, Pitetti K, Agiovlasitis S, Guerra-Junior G. Overweight and obesity in children and adolescents with Down syndrome-prevalence, determinants, consequences, and interventions: A literature review. Res Dev Disabil. 2016 Oct;57:181-92. doi: 10.1016/j.ridd.2016.06.018. Epub 2016 Jul 19. PMID 27448331
- [Background] Pecoraro L, Ferron E, Solfa M, Mirandola M, Lauriola S, Piacentini G, Pietrobelli A. Body composition and laboratory parameters in children with down syndrome: The DONUT study. Clin Nutr ESPEN. 2023 Oct;57:253-257. doi: 10.1016/j.clnesp.2023.07.003. Epub 2023 Jul 10. PMID 37739665
- See also: Related Info — https://ensati.wixsite.com/ensati